CLINICAL TRIAL: NCT03091465
Title: Validation of the International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) Prognostic Classification for Targeted Therapies (TKI/mTOR Inhibitors) in Second Line After First Line Treatment With Pazopanib
Acronym: Spazo-2
Status: Completed | Type: Observational
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Other Study IDs: SOGUG-2016-A-IEC(REN)-4; SOG-PAZ-2016-01 (Other: The Spanish Agency of Medicinal Products and Medical Devices)
Record Dates: First submitted 2017-03-02; First posted 2017-03-27 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic Renal Cell Carcinoma patients: This is a nation-wide retrospective observational study with patients treated with first-line pazopanib for mRCC in daily clinical practice since April 2011 (date of approval of pazopanib in Spain), January 2016.

SUMMARY:
This is a nation-wide retrospective observational study which will be performed in 50 centres in Spain, geographically representative of all regions, with at least 5 patients treated with first-line pazopanib for mRCC in daily clinical practice since April 2011 (date of approval of pazopanib in Spain), January 2016.

Pazopanib is one of the standard tyrosine-kinase inhibitors (TKI) for the first-line treatment of metastatic renal cell carcinoma. In our previous SPAZO study, the Spanish Oncologic Genitourinary Group (SOGUG) validated the IMDC prognostic classification for patients receiving first-line pazopanib, and demonstrated the effectiveness of this drug in routine clinical practice. However, in this series of 278 patients, we could not obtain enough information on the effectiveness of pazopanib in special subpopulations such as non-clear cell histologies, and others subgroups, due to a small simple size of each of these subpopulations. On the other hand, after the results of RECORD-1 and AXIS trials, switching to everolimus or axitinib is the current approach for patients who progresses to a first-line TKI. However, these pivotal studies did not include patients treated with first-line pazopanib study because this drug was not available at that time. The results of the SPAZO study also suggested that the effectiveness of second-line targeted therapies (TT) after pazopanib in routine clinical practice is similar to the observed in clinical trials after sunitinib, sorafenib or bevacizumab. In addition, the preliminary results indicated that there are not meaningful differences in the effectiveness of TKI or mTOR inhibitors after pazopanib, when the results are adjusted by the IMDC prognostic classification. However, the IMDC prognostic classification for second-line TT has not yet been validated for patients who receive pazopanib as first-line. In addition our sample size was not large enough to make a comparison of effectiveness between mTOR inhibitors and antiVEGF for each prognostic subgroups of the IMDC.

Based on that, the Spanish Oncologic Genitourinary Group has decided to launch the SPAZO-2 study, in which we intend to prolong the follow up of patients included in SPAZO, and to increase the sample size with new patients from new centres, in order to obtain a larger sample in each of the subpopulations of interest, with the objective of obtaining more information about the above questions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with confirmed mRCC. All histologies are allowed.
* 2. Patients who have received pazopanib in their centre as first TKI for metastatic renal carcinoma in daily clinical practice since its approval in Spain until January 2016 (previous non-TKI therapies such as surgery for metastasis, local radiotherapy, citokines or chemotherapy are allowed.
* 3. Age ≥18 years.
* 4. Patients alive should give informed consent to participate in the study and to allow their medical records to be reviewed, preferably in writing o orally before independent witnesses of the research team and after being informed and have sufficient time to decide on their inclusion in the study

Exclusion Criteria:

* 1. Patients who received pazopanib in any clinical trial, or who had received any systemic therapy prior to pazopanib will not be included, except citoquines or sunitinib providing it had been given as first-line, and switched to pazopanib due to toxicity or intolerance during the first cycle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic renal cell carcinoma patients treated with pazopanib as first line treatment and target therapies (TKI/mTOR inhibitors) in second line
Sampling Method: Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

PRIMARY OUTCOMES:
IMDC prognostic | 1 day
  Validate the IMDC prognostic classification in terms of overall survival, for second line treatment with mTOR/TKI inhibitors after first-line pazopanib. Overall survival defined as the period between second-line targeted therapy initiation and the date of death or censored on the day of last follow up visit, will be indirectly compared to the reported in the IMDC for the overall population and for each IMDC subgroups.

SECONDARY OUTCOMES:
Effectiveness of mTOR inhibitors versus antiangiogenic TKI inhibitors in second-line after progression to pazopanib in the first-line setting of mRCC patients in terms of overall survival (OS). | 1 day
Effectiveness of mTOR inhibitors versus antiangiogenic TKI inhibitors in second-line after progression to pazopanib in the first-line setting of mRCC patients in terms of progression-free survival (PFS). | 1 day
Effectiveness of mTOR inhibitors versus antiangiogenic TKI inhibitors in second-line after progression to pazopanib in the first-line setting of mRCC patients in terms of response rate (RR). | 1 day
Effectiveness of pazopanib administered in the first-line setting of mRCC patients in terms of OS. | 1 day
Effectiveness of pazopanib administered in the first-line setting of mRCC patients in terms of PFS. | 1 day
Effectiveness of pazopanib administered in the first-line setting of mRCC patients in terms of RR. | 1 day
Safety of pazopanib and mTOR/TKI inhibitors evaluated as the number of patients who present treatment-related adverse events as assessed by CTCAE v4.0. | 1 day

CONTACTS AND LOCATIONS:
Locations (57):
- Spain (57):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Mútua Terrassa, Terrassa, Barcelona
  - Onkologikoa, Donostia / San Sebastian, Guipúzcoa
  - Complejo Hospitalario de Jaén, Jaén, Jaén
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de León, León, León
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Quirón, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital de Son Llàtzer, Palma de Mallorca, Mallorca
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Complexo Hospitalario Universitario de Ourense, Ourense, Ourense
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Universitario de La Ribera, Alzira, Valencia
  - Hospital de Basurto, Bilbao, Vizcaya
  - Clínica IMQ Zorrotzaurre, Bilbao, Vizcaya
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Juan Ramón Jimenez, Huelva
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital La Luz, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Central de la Defensa "Gómez-Ulla", Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Provincial de Pontevedra, Pontevedra
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Virgen del Rocío, Seville
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital Virgen de la Salud, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clinico de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario y Politécnico de La Fe, Valencia
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Result] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Result] Rini BI, Campbell SC, Escudier B. Renal cell carcinoma. Lancet. 2009 Mar 28;373(9669):1119-32. doi: 10.1016/S0140-6736(09)60229-4. Epub 2009 Mar 5. PMID 19269025